CLINICAL TRIAL: NCT04255342
Title: Clinical, Radiographic, and Histomorphometric Analysis of AstraTech Implant EV Placed and Immediately Provisionalized Into Preserved Alveolar Ridges: A Prospective 3-Year Outcomes Study
Brief Title: Azento IIS 3 Year Outcomes Implant Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and PI mutual agreement to discontinue study early due to change in statistical analysis of data.
Sponsor: Christopher Barwacz (Other)
Responsible Party: Sponsor-Investigator, Christopher Barwacz, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201911024
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Tooth Loss
Keywords: alveolar bone; alveolar ridge; bone grafting; bone resorption; dental implant
MeSH Terms: conditions — Tooth Loss; Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Implant Placement and Temporary Crown using AstraTech Implant System EV, Final Crown Delivery (Experimental)
  Interventions: Device: Implant Placement and Temporary Crown using AstraTech Implant System EV, Final Crown Delivery

INTERVENTIONS:
Device: Implant Placement and Temporary Crown using AstraTech Implant System EV, Final Crown Delivery — At least 3 months after tooth removal and bone grafting, a dental implant will be placed using Azento, a commercially-available product that uses computer technology to plan the dental implant placement using the AstraTech Implant System EV and an immediate implant temporary crown using Azento. After 3 months with the temporary crown, a definitive all-ceramic crown, made using a digital workflow will be placed.

SUMMARY:
The revised purpose of this study is to compare and evaluate the stability of the implant body, survival rate, bone-level changes, and the implant's soft-tissue outcomes over a period of 1 year. Only 1 tooth is studied per participant.

In July of 2024, the revised protocol and revised Statistical Analysis plan were amended post-hoc, and the revised protocol and statistical analysis plan were approved by the IRB review committee in July of 2024.

As a result, the study has been terminated due to a change in the study's data analysis, and so the study will only analyze data up to and including the 1-year point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may identify as either male, female, or intersex
* Age: 18 years or older
* Subjects with a healed, single-rooted tooth (except mandibular incisors) that has previously undergone ARP-SG with particulate allograft material within the past 2 months.
* Subjects must have stable occlusion, with absence of caries or other known acute pathology (i.e., untreated endodontic lesion, periodontal abscess, external/internal resorption, etc.) on teeth proximal to the implant site that would negatively influence implant outcomes
* Must be in adequate physical and mental health to undergo routine dental treatment including the surgical procedures associated tooth extraction and implant placement
* Subjects' treatment plan must include replacement of the tooth to be extracted with dental implant supported fixed restoration
* Subjects must have read, understood and signed an informed consent form
* Subjects must be willing to return for the required number of visits
* Subjects' tooth must be a permanent tooth, not a primary tooth (also known as baby tooth).

Exclusion Criteria:

* Mandibular incisors
* Acute infection associated with the tooth to be extracted or with adjacent teeth
* Unstable occlusion, presence of caries or other acute pathology on teeth adjacent to the implant site
* History of significant heart, stomach, liver, kidney, blood, immune system disease, or other organ impairment or systemic diseases that would prevent undergoing the proposed treatment or may result in compromised healing (e.g. poorly controlled diabetes, active heavy tobacco use [>10 cigs/day]), history of head/neck radiation, history of chemotherapy within the last 5 years
* Subjects with uncontrolled and/or severe metabolic bone diseases or disorders, such as osteoporosis, thyroid disorders or Paget's disease
* Subjects taking any medication or supplement known to largely influence bone metabolism, such as IV bisphosphonates, long-term history of oral bisphosphonates or chronic intake of glucocorticoids
* Pregnant women or nursing mothers
* Subjects that are unwilling or unable to sign the informed consent
* History of lack of compliance with dental visits
* Subjects unwilling to return for the required number of visits
* Subject currently undergoing orthodontic treatment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barwacz, DDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alkan EA, Parlar A, Yildirim B, Senguven B. Histological comparison of healing following tooth extraction with ridge preservation using enamel matrix derivatives versus Bio-Oss Collagen: a pilot study. Int J Oral Maxillofac Surg. 2013 Dec;42(12):1522-8. doi: 10.1016/j.ijom.2013.06.002. Epub 2013 Jul 8. PMID 23845297
- [Background] Araujo M, Linder E, Wennstrom J, Lindhe J. The influence of Bio-Oss Collagen on healing of an extraction socket: an experimental study in the dog. Int J Periodontics Restorative Dent. 2008 Apr;28(2):123-35. PMID 18546808
- [Background] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Background] Araujo MG, Liljenberg B, Lindhe J. Dynamics of Bio-Oss Collagen incorporation in fresh extraction wounds: an experimental study in the dog. Clin Oral Implants Res. 2010 Jan;21(1):55-64. doi: 10.1111/j.1600-0501.2009.01854.x. PMID 20070748
- [Background] Arora H, Khzam N, Roberts D, Bruce WL, Ivanovski S. Immediate implant placement and restoration in the anterior maxilla: Tissue dimensional changes after 2-5 year follow up. Clin Implant Dent Relat Res. 2017 Aug;19(4):694-702. doi: 10.1111/cid.12487. Epub 2017 Apr 21. PMID 28429394
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Barwacz, C. & Hernandez, M. (2013) Maximizing Esthetics of Fixed Interim Restorations via Direct Extrinsic Characterization. Journal of Cosmetic Dentistry 29, 122-131.
- [Background] Barwacz CA, Pantzlaff E, Allareddy V, Avila-Ortiz G. Graduate Periodontics Programs' Integration of Implant Provisionalization in Core Curricula: Implementation of CODA Standard 4-10.2.d. J Dent Educ. 2017 Jun;81(6):696-706. doi: 10.21815/JDE.016.033. PMID 28572416
- [Background] Barwacz CA, Stanford CM, Diehl UA, Cooper LF, Feine J, McGuire M, Scheyer ET. Pink Esthetic Score Outcomes Around Three Implant-Abutment Configurations: 3-Year Results. Int J Oral Maxillofac Implants. 2018 Sep/Oct;33(5):1126-1135. doi: 10.11607/jomi.6659. PMID 30231101
- [Background] Cooper LF, Reside G, Stanford C, Barwacz C, Feine J, Nader SA, Scheyer T, McGuire M. Three-Year Prospective Randomized Comparative Assessment of Anterior Maxillary Single Implants with Different Abutment Interfaces. Int J Oral Maxillofac Implants. 2019 Jan/Feb;34(1):150-158. doi: 10.11607/jomi.6810. PMID 30695089
- [Background] Cooper LF, Tarnow D, Froum S, Moriarty J, De Kok IJ. Comparison of Marginal Bone Changes with Internal Conus and External Hexagon Design Implant Systems: A Prospective, Randomized Study. Int J Periodontics Restorative Dent. 2016 Sep-Oct;36(5):631-42. doi: 10.11607/prd.2433. PMID 27560668
- [Background] Crespi R, Cappare P, Crespi G, Gastaldi G, Romanos GE, Gherlone E. Tissue Remodeling in Immediate Versus Delayed Prosthetic Restoration in Fresh Socket Implants in the Esthetic Zone: Four-Year Follow-up. Int J Periodontics Restorative Dent. 2018;38(Suppl):s97-s103. doi: 10.11607/prd.3123. Epub 2018 Mar 7. PMID 29513776
- [Background] De Rouck T, Collys K, Wyn I, Cosyn J. Instant provisionalization of immediate single-tooth implants is essential to optimize esthetic treatment outcome. Clin Oral Implants Res. 2009 Jun;20(6):566-70. doi: 10.1111/j.1600-0501.2008.01674.x. Epub 2009 Mar 3. PMID 19302238
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Heberer S, Al-Chawaf B, Hildebrand D, Nelson JJ, Nelson K. Histomorphometric analysis of extraction sockets augmented with Bio-Oss Collagen after a 6-week healing period: a prospective study. Clin Oral Implants Res. 2008 Dec;19(12):1219-25. doi: 10.1111/j.1600-0501.2008.01617.x. No abstract available. PMID 19040436
- [Background] Heinemann F, Hasan I, Schwahn C, Bourauel C, Mundt T. Bone level change of extraction sockets with Bio-Oss collagen and implant placement: a clinical study. Ann Anat. 2012 Nov;194(6):508-12. doi: 10.1016/j.aanat.2011.11.012. Epub 2011 Dec 23. PMID 22244384
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Kan JY, Rungcharassaeng K, Lozada J. Immediate placement and provisionalization of maxillary anterior single implants: 1-year prospective study. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):31-9. PMID 12608666
- [Background] Kan JY, Rungcharassaeng K, Umezu K, Kois JC. Dimensions of peri-implant mucosa: an evaluation of maxillary anterior single implants in humans. J Periodontol. 2003 Apr;74(4):557-62. doi: 10.1902/jop.2003.74.4.557. PMID 12747463
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Nart J, Barallat L, Jimenez D, Mestres J, Gomez A, Carrasco MA, Violant D, Ruiz-Magaz V. Radiographic and histological evaluation of deproteinized bovine bone mineral vs. deproteinized bovine bone mineral with 10% collagen in ridge preservation. A randomized controlled clinical trial. Clin Oral Implants Res. 2017 Jul;28(7):840-848. doi: 10.1111/clr.12889. Epub 2016 Jun 22. PMID 27335267
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Noelken R, Oberhansl F, Kunkel M, Wagner W. Immediately provisionalized OsseoSpeed() Profile implants inserted into extraction sockets: 3-year results. Clin Oral Implants Res. 2016 Jun;27(6):744-9. doi: 10.1111/clr.12651. Epub 2015 Aug 24. PMID 26300062
- [Background] Ponsi J, Lahti S, Rissanen H, Oikarinen K. Change in subjective oral health after single dental implant treatment. Int J Oral Maxillofac Implants. 2011 May-Jun;26(3):571-7. PMID 21691604
- [Background] Raes F, Cooper LF, Tarrida LG, Vandromme H, De Bruyn H. A case-control study assessing oral-health-related quality of life after immediately loaded single implants in healed alveolar ridges or extraction sockets. Clin Oral Implants Res. 2012 May;23(5):602-8. doi: 10.1111/j.1600-0501.2011.02178.x. Epub 2011 Apr 19. PMID 21504481
- [Background] Roccuzzo M, Gaudioso L, Lungo M, Dalmasso P. Surgical therapy of single peri-implantitis intrabony defects, by means of deproteinized bovine bone mineral with 10% collagen. J Clin Periodontol. 2016 Mar;43(3):311-8. doi: 10.1111/jcpe.12516. Epub 2016 Mar 9. PMID 26800389
- [Background] Scheyer ET, Heard R, Janakievski J, Mandelaris G, Nevins ML, Pickering SR, Richardson CR, Pope B, Toback G, Velasquez D, Nagursky H. A randomized, controlled, multicentre clinical trial of post-extraction alveolar ridge preservation. J Clin Periodontol. 2016 Dec;43(12):1188-1199. doi: 10.1111/jcpe.12623. Epub 2016 Oct 21. PMID 27617409
- [Background] Spyropoulou PE, Razzoog M, Sierraalta M. Restoring implants in the esthetic zone after sculpting and capturing the periimplant tissues in rest position: a clinical report. J Prosthet Dent. 2009 Dec;102(6):345-7. doi: 10.1016/S0022-3913(09)60189-X. PMID 19961991
- [Background] Stanford CM, Barwacz C, Raes S, De Bruyn H, Cecchinato D, Bittner N, Brandt J. Multicenter Clinical Randomized Controlled Trial Evaluation of an Implant System Designed for Enhanced Primary Stability. Int J Oral Maxillofac Implants. 2016 Jul-Aug;31(4):906-15. doi: 10.11607/jomi.4869. PMID 27447160
- [Background] Strietzel FP, Neumann K, Hertel M. Impact of platform switching on marginal peri-implant bone-level changes. A systematic review and meta-analysis. Clin Oral Implants Res. 2015 Mar;26(3):342-58. doi: 10.1111/clr.12339. Epub 2014 Jan 20. PMID 24438506
- [Background] Su H, Gonzalez-Martin O, Weisgold A, Lee E. Considerations of implant abutment and crown contour: critical contour and subcritical contour. Int J Periodontics Restorative Dent. 2010 Aug;30(4):335-43. PMID 20664835

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implant Placement and Temporary Crown Using AstraTech Implant System EV, Final Crown Delivery
Started | 25
Completed | 22
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population differs from the final results, because 3 subjects were lost to follow-up over the course of the study.
Arm/Group | Implant Placement and Temporary Crown Using AstraTech Implant System EV, Final Crown Delivery
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Had an Implant That Survived 1 Year After Permanent Final Crown Placement.
Description: For participants that had permanent restoration of the final crown performed, this outcome is determined via clinical evaluation of the percentage of participants that still had their 1 implant in place after 1 year of having the permanent final crown placement. Note: Only 1 implant was placed per participant.
Time Frame: 1 year after permanent final crown placement
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Placement and Temporary Crown Using AstraTech Implant System EV, Final Crown Delivery
Number analyzed (Participants) | 22
Participants | 22

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Implant Placement and Temporary Crown Using AstraTech Implant System EV, Final Crown Delivery
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT04255342/Prot_SAP_000.pdf